CLINICAL TRIAL: NCT03191682
Title: A Phase I, First-in-Human Study of PRL3-ZUMAB In Advanced, Solid Tumors and Haematologic Malignancies
Brief Title: A First-in-Human Study of PRL3-ZUMAB
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: INTRA-IMMUSG PRIVATE LIMITED (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC03/06/16
Record Dates: First submitted 2017-02-13; First posted 2017-06-19 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PRL3-ZUMAB (Experimental): The starting dose will be 0.3 mg/kg, administered Q2 weekly, with the subsequent dose levels being 0.9 mg/kg, 3.0 mg/kg, and 6.0 mg/kg, all administered on a Q2 weekly basis until disease progression
  Interventions: Drug: PRL3-ZUMAB

INTERVENTIONS:
Drug: PRL3-ZUMAB — The starting dose will be 0.3 mg/kg, administered Q2 weekly, with the subsequent dose levels being 0.9 mg/kg, 3.0 mg/kg, and 6.0 mg/kg, all administered on a Q2 weekly basis until disease progression. The investigator will monitor each subject for the occurrence of AEs. In event of infusion-related adverse events, the Investigator, in consultation with the PI, may increase the duration of the infusion over a period of up to 24 hours at their discretion. Dosing will continue in a standard 3+3 design for dose escalation.

SUMMARY:
This study is carried out to test the safety of a study drug called PRL3-ZUMAB. PRL3-ZUMAB is an investigational drug that has not yet been approved by the Food and Drug Administration (FDA) or any other regulatory authorities for commercial purposes. This is the first study in which PRL3-ZUMAB will be given to humans. The study drug has been tested in animals and was found to be well-tolerated with minimal side effects. This research study will test different doses of the drug to see which dose is safest in people.

DETAILED DESCRIPTION:
PRL-3 is involved in cellular processes driving metastasis, including cell proliferation, invasion, motility and survival and has been shown to be upregulated and overexpressed in cancer tissues, in contrast to low or no expression in most normal tissues. In mouse models of PRL3-positive gastric cancers, PRL3-ZUMAB, a first-in-class humanized antibody against PRL-3, has shown to reduce tumour growth and increase survival. In contrast, no response was seen in PRL3-negative gastric cancer mouse models, reflecting the exquisite target specificity of PRL3-ZUMAB.

Because PRL3-ZUMAB has produced little apparent toxicity in Good Laboratory Practice (GLP) toxicology studies, it is expected to have a favorable adverse event (AE) profile in humans. PRL3-ZUMAB has the potential to be an anti-tumor agent in the management of solid tumors. In this first-in-human study, the Phase Ia study will confirm safety, tolerability and establish evidence for anti-tumor activity in advanced, solid tumor patients in the dose expansion phase (Phase Ib).

- Rationale for Doses Selected: Administration of 50-150 μg PRL3-zumab/dose significantly reduced PRL-3-positive lung tumor burden in Balb/C nude mice metastatic tumor models (p = 0.044, Kruskal-Wallis test).

These results established the range of 50-150 ug PRL3-zumab/dose as sufficiently efficacious exposure levels for maximal suppression of PRL-3-positive tumors in rodents in this experimental setting. Importantly, this dose range did not cause any undesirable side effects - mice receiving these doses of PRL3-zumab displayed normal weight gain and physical activity, as compared to untreated mice. Based on these observations, the median dose of 100 ug PRL3-zumab/dose (i.e. approximately 4-5 mg/kg, depending on mice body weight between 20 to 25 g) was set as the pharmacologically active dose (PAD) in all subsequent animal treatment experiments. Assuming a PAD in rodent tumor models of 5 mg/kg, a PAD of around 0.4 mg/kg is expected in humans by converting this into the Minimal Anticipated Biologically Effect Level (MABEL) in humans by dividing by a factor of 12.3 (based on FDA Guidance for Industry: Estimating the Maximum Safe Starting Dose in Initial Clinical Trials for Therapeutics in Adult Healthy Volunteers).

In the monkey toxicokinetics study, PRL3-zumab was administered IV over 8 weeks at 2 week intervals. Dose amounts of 4 to 36 mg/kg (0 mg/kg for controls) were used. As the dose increased from 4 to 36 mg/kg, the systemic exposure (AUC0-168 and C0) to PRL3-zumab increased dose-proportionally on Day 1 and 57 and there was no marked drug accumulation for PRL3-zumab at any dose level. Therefore, the no observed adverse effect level (NOAEL) in the GLP toxicology study in cynomolgus monkeys for PRL3-zumab was considered to be 36 mg/kg/dose.

Using the standard safety factor of 1/10th of the NOAEL as the starting dose for humans yields a human dose of 3.6 mg/kg/dose. As this is a first-in-class compound and first-in-human study, the investigators have factored in a greater safety margin of an additional 1/10th of the starting dose,resulting in a final starting dose of 0.3 mg/kg/dose. Importantly, while this starting dose provides a 100-fold safety margin compared to the NOAEL, it is also within the estimated human PAD range (as determined from rodent studies).

The investigators will perform 3-fold escalations from 0.3 mg/kg to 6 mg/kg and will use the correlative PK and PDn data to guide further doses and to determine the maximum tolerated dose (MTD) and optimum biologic dose (OBD).

Taking into account the pharmacologically active dose (PAD) in mouse tumor models of 5 mg/kg, and converting this into the human effective dose (HED) by a factor of 12.3 (based on FDA Guidance for Industry: Estimating the Maximum Safe Starting Dose in Initial Clinical Trials for Therapeutics in Adult Healthy Volunteers), a PAD of 0.4 mg/kg is expected for humans. Thus, the proposed final starting dose of 0.3 mg/kg/dose is indeed within the PAD range.

Before the start of each new dose cohort, a review of the adverse event profile and pharmacokinetics (where available) will be conducted by the investigators before dose escalation.

Once the MTD or OBD has been determined, the investigators will conduct the dose expansion part (phase Ib) of the study which will include PRL3-positive tumors.

- Rationale for Study Population: As this is a FIH study, the risk-benefit ratio of the drug is unknown. Therefore, the study population of patients with advanced solid tumors who no longer respond to standard therapy or for whom no standard therapy is available, would be appropriate for this study as they may benefit from treatment with PRL3-ZUMAB.

- Rationale for Study Design: This phase 1, open label, dose-escalation study of PRL3-ZUMAB will use titration from low doses to higher doses of PRL3-ZUMAB in order to assess the PK, PDn, and potential toxicities of the study drug in the target population, and to determine the MTD/OBD/ or recommended phase 2 dose (RP2D). The sample size employed is a minimally modified standard 3+3 cohort model commonly used in Phase I oncology studies. Once determined, the MTD/OBD/RP2D may be administered to an Expansion Cohort (Phase Ib) of subjects with advanced PRL-3 expressing cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent. Written informed consent must be obtained prior to performing any study-related procedures.
2. Histopathological- or cytological- documented, measurable or non-measurable, locally advanced unresectable primary or metastatic solid tumor unresponsive to standard therapy or for which there is no standard therapy available.
3. Progressive disease (PD) during or following the last treatment regimen as defined by the Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v 1.1 guidelines)
4. Haematologic malignancies study population for expansion cohort:

   * Newly diagnosed early AML (age>65 years) who are unfit for the intensive chemotherapy and declined hypomethylating agent
   * Elderly AML who failed first line of treatment including hypomethylating agent
   * Relapsed or refractory AML who failed at least 1 line of salvage chemotherapy and are deemed unfit for further intensive chemotherapy
   * Relapsed or refractory multiple myeloma who failed at least 3 lines of prior therapy and with measurable disease either by serum M-protein, involved immunoglobulin type or serum free light chain.
5. Life expectancy >3 months
6. Eastern Cooperative Oncology Group (ECOG) performance status (ECOG PS) score of <= 2 at study entry
7. Age ≥ 21 years
8. Pre-study echocardiogram or multigated acquisition (MUGA) scan with left ventricular ejection fraction (LVEF) ≥ 50%
9. Recovery to Grade ≤ 1 by the Common Terminology Criteria for Adverse Events, Version 4.03 (CTCAE v 4.03), from the effects of recent surgery, radiotherapy, chemotherapy, hormonal therapy, or other targeted therapies for cancer, with the exception of alopecia or peripheral neuropathy (the latter of which must have resolved to Grade ≤ 2).
10. Women of childbearing potential (WOCBP) must have a negative pregnancy test at study entry. Subjects not considered WOCBP are those without menses for 24 consecutive months, and those who have undergone hysterectomy and/or bilateral salpingo-oophorectomy. WOCBP must be willing to use acceptable methods of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, or condom with spermicide, or abstinence) for the duration of the study.
11. Preserved organ function as defined below. All parameters must be evaluated within 7 days prior to the first dose of PRL3-ZUMAB:

    * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 X upper limit of normal (ULN), or ≤ 5.0 X ULN in subjects with metastatic liver disease
    * Hemoglobin ≥ 9 g/dL
    * Total bilirubin ≤ 1.5 × ULN
    * Creatinine ≤ 1.5 × ULN
    * Absolute neutrophil count (ANC) ≥ 1.5 × 109/L (only applicable to non-AML subject)
    * Platelets ≥ 100 × 109/L (only applicable to non-AML subject)

Exclusion Criteria:

1. Prior anti-cancer chemotherapy, hormonal therapy, radiotherapy, immunotherapy, monoclonal antibodies, targeted therapy or investigational agents within 4 weeks (6 weeks for mitomycin C and nitrosoureas) prior to the first dose of PRL3-ZUMAB
2. Known symptomatic brain metastases. Subjects with treated brain metastasis (radiotherapy and/or surgery) will be eligible if they:

   * Have completed treatment for their brain metastasis > 4 weeks prior to scheduled study treatment start date;
   * Are neurologically stable;
   * Are not receiving corticosteroids or corticosteroids in doses no greater than physiological replacement (e.g., dexamethasone < 1.5 mg/day); and
   * Have a screening/baseline MRI scan of the brain that specifically verifies no evidence of CNS hemorrhage and no active gadolinium enhancing lesions.
3. Isolated CNS disease in AML cohort
4. Acute promyelocytic leukemia or AML M3
5. Non-secretary myeloma
6. Primary brain / CNS malignancy (e.g., gliomas, lymphomas)
7. Leptomeningeal disease
8. Pregnancy (confirmed by beta -human chorionicgonadotrophin [β-HCG] or lactating
9. Significant uncontrolled intercurrent illness including, but not limited to:

   * ongoing or active infection requiring parenteral antibiotics; clinically significant cardiac disease [(class II, III, or IV of the New York Heart Association classification (NYHA)];
   * unstable angina pectoris, myocardial infarction within 6 months or is post angioplasty or stenting within 6 months;
   * uncontrolled hypertension (i.e., systolic blood pressure (BP) > 150 mm Hg, diastolic BP > 90 mm Hg), found on two consecutive measurements separated by a 1-week period;
   * clinically significant cardiac arrhythmia; or
   * uncontrolled diabetes.
10. Known human immunodeficiency virus infection or acquired immunodeficiency syndrome-related illness
11. Known active hepatitis B or C or other active (nonmalignant) liver disease. Patients with hepatitis B surface antigen positive serology may participate if HBV DNA copy number is <100 copies/mL.
12. History of previously treated neurologic or other neurodegenerative diseases/disorders, or psychiatric illness, disability, or social situation that would compromise the subject's safety, ability to provide consent, or limit his/her compliance with study requirements
13. Prior hypersensitivity reaction to monoclonal antibodies or other therapeutic proteins, and the reaction could not be controlled or prevented on subsequent infusion with standard therapies such as antihistamines, 5-HT3 antagonists, or corticosteroids.
14. History of another primary cancer, with the exception of:

    * curatively resected nonmelanomatous skin cancer,
    * curatively treated cervical carcinoma in-situ,
    * prostate cancer treated with leuteinizing hormone-releasing hormone (LH-RH) agonists/pure antagonists for at least 2 months, or
    * other primary solid tumor treated with curative intent and no known active disease present and no treatment administered during the last 3 years.
15. Require treatment with prohibited concomitant medications
16. Prior stem cell or bone marrow transplant
17. Vaccinated within 8 weeks from prior to the first administration of PRL3-ZUMAB

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2017-02-20 (Actual); Primary Completion 2027-02-20 (Estimated); Study Completion 2027-02-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of Grade 3 or 4 drug related adverse events and clinical lab abnormalities defined as Dose Limiting Toxicities (DLTs) using NCI CTCAE v 4.03 | During cycle 1 (28 days) of treatment
Maximum tolerated dose of PRL3-zumab, defined as the highest dose level at which < 33% of 6 patients experience a dose-limiting toxicity graded according to Common Terminology Criteria for Adverse Events version 4 (Phase I) | 28 days
Recommended Phase 2 Dose (RP2D) of PRL3-zumab defined as the most appropriate dose to maximize a favorable risk/benefit reward for the participant population | After completion of all Cycle 1 (28 days) of treatment for participant enrolled in part 1

SECONDARY OUTCOMES:
Total Active Pharmaceutical Ingredient (API) levels in plasma | The pharmacokinetics profile will be assessed by blood collection during Cycle 1 (28 days) of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Cheng Ean Chee, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zeng Q, Hong W, Tan YH. Mouse PRL-2 and PRL-3, two potentially prenylated protein tyrosine phosphatases homologous to PRL-1. Biochem Biophys Res Commun. 1998 Mar 17;244(2):421-7. doi: 10.1006/bbrc.1998.8291. PMID 9514946
- [Background] Al-Aidaroos AQ, Zeng Q. PRL-3 phosphatase and cancer metastasis. J Cell Biochem. 2010 Dec 1;111(5):1087-98. doi: 10.1002/jcb.22913. PMID 21053359
- [Background] Walls CD, Iliuk A, Bai Y, Wang M, Tao WA, Zhang ZY. Phosphatase of regenerating liver 3 (PRL3) provokes a tyrosine phosphoproteome to drive prometastatic signal transduction. Mol Cell Proteomics. 2013 Dec;12(12):3759-77. doi: 10.1074/mcp.M113.028886. Epub 2013 Sep 12. PMID 24030100
- [Derived] Chee CE, Ooi M, Lee SC, Sundar R, Heong V, Yong WP, Ng CH, Wong A, Lim JSJ, Tan DSP, Soo R, Tan JTC, Yang S, Thura M, Al-Aidaroos AQ, Chng WJ, Zeng Q, Goh BC. A Phase I, First-in-Human Study of PRL3-zumab in Advanced, Refractory Solid Tumors and Hematological Malignancies. Target Oncol. 2023 May;18(3):391-402. doi: 10.1007/s11523-023-00962-w. Epub 2023 Apr 15. PMID 37060431